CLINICAL TRIAL: NCT03265028
Title: National Implementation of a Multifaceted Web-based Communication Training to Reduce of Inappropriate Antibiotic Prescribing for (Lower) Respiratory Tract Infections
Brief Title: TRACE E-learning Implementation in Belgium
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Belgian Antibiotic Policy Coordination Committee (BAPCOC) (Unknown)
Responsible Party: Principal Investigator, Niels Adriaenssens, Dr., Universiteit Antwerpen
Other Study IDs: TRACE Implementation
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Respiratory Tract Infections
Keywords: primary care; antibiotics; communication skills; general practice; outpatient; ambulatory care; anti-bacterial agents
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention: Invited to take the TRACE e-learning.
  Interventions: Behavioral: TRACE e-learning
- Control: Not (yet) invited to take the TRACE e-learning.

INTERVENTIONS:
Behavioral: TRACE e-learning — The TRACE e-learning (www.acutecough.org) is an educational web-based module including communication training for physicians, and includes patient booklets to be used interactively during the consultation.
  Groups: Intervention

SUMMARY:
Antibiotic resistance is a worldwide health care problem. Increasing use of antibiotics is associated with an increase in the prevalence of bacteria resistant to the antibiotic used. Reducing antibiotic use can be effected by improving antibiotic prescribing quality in two complementary ways. One is to limit antibiotic prescribing to those patients who will benefit from the treatment and two is to prescribe these patients the recommended antibiotic.

International research has shown that a web-based communication training for the prescriber combined with an interactive booklet containing relevant patient information (Genomics to combat Resistance against Antibiotics for Community acquired LRTI in Europe INternet Training for Reducing antibiOtic use (GRACE INTRO)) can significantly and safely reduce antibiotic prescribing in adults presenting to primary care with acute cough/lower respiratory tract infections (LRTI). Quality assessment of antibiotic prescribing for respiratory infections in general practice has revealed the use of far too many (broad-spectrum) antibiotics in Belgium.

In the proposed project, the investigators aspire to make Belgium the first European country to implement the most cost-effective part of the GRACE INTRO intervention (Translational Research on Antimicrobial resistance and Community-acquired infections in Europe (TRACE) e-learning, www.acutecough.org) at national level and to perform a scientifically sound assessment of the nationwide implementation on outpatient antibiotic use and societal cost.

DETAILED DESCRIPTION:
The envisaged research aims to implement the most cost-effective part of the GRACE INTRO intervention (TRACE e-learning, www.acutecough.org), i.e. a web-based communication training and an interactive patient booklet for adults presenting to primary care with LRTI, at national level. For that purpose the investigators will perform a stepped wedge cluster-randomised trial. Stepped wedge randomised trial designs involve sequential roll-out of an intervention to participants (individuals or clusters) over a number of time periods. By the end of the study, all participants will have received the intervention, although the order in which participants receive the intervention is determined at random. Over a period of one year all practices in the 10 Belgian provinces and Brussels (n=11 clusters) will get access to the intervention. The order in which the clusters receive the intervention is determined at random. The general practitioners (GPs) in the intervention phase will be invited to take an educational web-based module, including communication training, to improve prescribing of antibiotics for LRTI and will receive patient booklets to be used interactively during the consultation. The clusters not yet exposed to the intervention will serve as control group. The effect on prescribing behavior will be assessed using monthly Intermutualistic Agency (IMA, www.nic-ima.be) data. Hence, the outcome measurement will have complete response, and will not interfere with the normal routine of the eligible GPs, allowing a more valid estimate of any intervention effect. Since the training will be assessed, and not the eligible practices or GPs, IMA has the legal authority (Art. 153 of the coordinated Law of 14 July 1994) to perform the required analyses. The estimates of the efficacy of the intervention will at the same time describe its effectiveness in daily practice, which is unconventional for a randomized trial (on a behavioural intervention). Given the large sample size, the proposed trial will also provide very precise estimates.

ELIGIBILITY:
Inclusion Criteria:

* all clinicians registered as General Practitioner in Belgium

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all clinicians registered as General Practitioner in Belgium
Sampling Method: Non-Probability Sample
Enrollment: 15802 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Antibiotic use (short term) | First 2 months after intervention
  Number of packages for antibacterials for systemic use (ATC J01) collected at the pharmacy (reimbursement data) per 1000 inhabitants per day

SECONDARY OUTCOMES:
Antibiotic use (intermediate term) | 3-6 months after intervention
  Number of packages for antibacterials for systemic use (ATC J01) collected at the pharmacy (reimbursement data) per 1000 inhabitants per day
Antibiotic use (long term) | 6-12 months after intervention
  Number of packages for antibacterials for systemic use (ATC J01) collected at the pharmacy (reimbursement data) per 1000 inhabitants per day

OTHER OUTCOMES:
Response rate (short term) | First 2 months after intervention
  The number of invited GPs taking the TRACE e-learning
Response rate (long term) | First year after intervention
  The number of invited GPs taking the TRACE e-learning

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Coenen, Prof, Principal Investigator — Universiteit Antwerpen
Locations (11):
- Belgium (11):
  - GPs of Henegouwen, Mons, Henegouwen
  - GPs of Limburg, Hasselt, Limburg
  - GPS of Luik, Liège, Luik
  - Gps of Luxemburg, Arlon, Luxemburg
  - GPs of Namen, Namur, Namen
  - GPs of Oost-Vlaanderen, Ghent, Oost-Vlaanderen
  - GPs of Vlaams-Brabant, Leuven, Vlaams-Brabant
  - GPs of Waals-Brabant, Wavre, Waals-Brabant
  - GPs of West-Vlaanderen, Bruges, West-Vlaanderen
  - GPs of Antwerp, Antwerp
  - GPs of Brussels, Brussels

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anthierens S, Tonkin-Crine S, Douglas E, Fernandez-Vandellos P, Krawczyk J, Llor C, Cals JW, Francis NA, Yardley L, Coenen S, Verheij T, Goossens H, Little P; GRACE INTRO study team. General practitioners' views on the acceptability and applicability of a web-based intervention to reduce antibiotic prescribing for acute cough in multiple European countries: a qualitative study prior to a randomised trial. BMC Fam Pract. 2012 Oct 11;13:101. doi: 10.1186/1471-2296-13-101. PMID 23110756
- [Background] Little P, Stuart B, Francis N, Douglas E, Tonkin-Crine S, Anthierens S, Cals JW, Melbye H, Santer M, Moore M, Coenen S, Butler C, Hood K, Kelly M, Godycki-Cwirko M, Mierzecki A, Torres A, Llor C, Davies M, Mullee M, O'Reilly G, van der Velden A, Geraghty AW, Goossens H, Verheij T, Yardley L; GRACE consortium. Effects of internet-based training on antibiotic prescribing rates for acute respiratory-tract infections: a multinational, cluster, randomised, factorial, controlled trial. Lancet. 2013 Oct 5;382(9899):1175-82. doi: 10.1016/S0140-6736(13)60994-0. Epub 2013 Jul 31. PMID 23915885
- [Background] Tonkin-Crine S, Anthierens S, Francis NA, Brugman C, Fernandez-Vandellos P, Krawczyk J, Llor C, Yardley L, Coenen S, Godycki-Cwirko M, Butler CC, Verheij TJ, Goossens H, Little P, Cals JW; GRACE INTRO team. Exploring patients' views of primary care consultations with contrasting interventions for acute cough: a six-country European qualitative study. NPJ Prim Care Respir Med. 2014 Jul 17;24:14026. doi: 10.1038/npjpcrm.2014.26. PMID 25030621
- [Background] Anthierens S, Tonkin-Crine S, Cals JW, Coenen S, Yardley L, Brookes-Howell L, Fernandez-Vandellos P, Krawczyk J, Godycki-Cwirko M, Llor C, Butler CC, Verheij T, Goossens H, Little P, Francis NA; GRACE/CHAMP INTRO team. Clinicians' views and experiences of interventions to enhance the quality of antibiotic prescribing for acute respiratory tract infections. J Gen Intern Med. 2015 Apr;30(4):408-16. doi: 10.1007/s11606-014-3076-6. Epub 2014 Nov 6. PMID 25373834
- [Derived] D'Hulster L, Abrams S, Bruyndonckx R, Anthierens S, Adriaenssens N, Butler CC, Verheij T, Goossens H, Little P, Coenen S. Nationwide implementation of online communication skills training to reduce overprescribing of antibiotics: a stepped-wedge cluster randomized trial in general practice. JAC Antimicrob Resist. 2022 Jun 29;4(3):dlac070. doi: 10.1093/jacamr/dlac070. eCollection 2022 Jun. PMID 35774072